CLINICAL TRIAL: NCT05696171
Title: Clinical Evaluation of Robot-assisted Cochlear Implant Insertion in Adults Using RobOtol® Compared to Manual Insertion
Acronym: ROBIICCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC22_0384
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Profound Bilateral Hearing Loss
Keywords: Profound hearing loss, cochlear implant, RobOtol®

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual insertion (Active Comparator): Manual insertion of the cochlear implant
  Interventions: Procedure: Cochlear implant manual insertion
- Robotized insertion (Experimental): Robotic insertion of the cochlear implant
  Interventions: Procedure: Cochlear implant robotized insertion

INTERVENTIONS:
Procedure: Cochlear implant manual insertion — Manual insertion of the cochlear implant into the round window during the surgery
  Arms: Manual insertion
Procedure: Cochlear implant robotized insertion — Robotic insertion of the cochlear implant into the round window during the surgery
  Arms: Robotized insertion

SUMMARY:
The purpose of this study is to evaluate, via a randomised controlled design, the efficacy of the robotic insertion of cochlear implant, versus manual insertion. Robotic insertion will be performed using Robotol.

This is a three years interventional study involving adults with profound bilateral hearing loss.

Eligible subjects will be randomized in two groups : robotic insertion, or manual insertion. Each patient will be followed during 12 months.

DETAILED DESCRIPTION:
Cochlear implants are currently the only option for the rehabilitation of bilateral profound hearing loss. Cochlear implant surgery efficacy has been largely demonstrated by numerous studies. But, despite multiple contributors, accuracy and sensitivity of cochlear implant insertion constitute the major and the single factor that surgeons have under control.

This manual surgery is performed in an extremely constrained environment and must be as much as delicate as possible to preserve patient's residual hearing potential. Manual insertion is still largely subject to experience and dexterity of the surgeon. Factors associated with the surgical insertion (such as incomplete or traumatic insertions, translocations, destruction of residual hearing) have a negative impact on final hearing correction performance.

To optimise the hearing results, the insertion must be precise, linear and atraumatic. These conditions may be achieved by robotic insertion.

The RobOtol® is an innovative robotic assistance system dedicated to ear surgery, designed and built in France. This is a compact serial robot with 7 degrees of freedom and high resolution, allowing lower insertion forces and higher insertion depth than the manual approach. Pilot clinical studies have already reported a reduced frequency of translocations via robotic assistance and a reduction in cochlear trauma.

The objective of Robiicca is to evaluate, via a randomised controlled design, the efficacy at 1 year of this robotic technology in cochlear implantation in adults.The hypothesis is that the optimization of the surgical procedure with the RobOtol® will maximize the audiometric results, as well as the residual hearing and the vestibular function.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age > 18)
* Eligible for a cochlear implant insertion according to the HAS recommendations
* Patient having signed an informed consent

Exclusion Criteria:

Exclusion Criteria:

* Profound hearing loss linked to meningitis
* Bilateral cochlear implants insertion during the same surgery
* Removal and re-insertion of a cochlear implant (due to a failure for example)
* Patient under guardianship or curatorship
* Contraindication to the use of the RobOtol®:

Patients wearing electronic devices directly connected to the brain or nervous system.

Presence of medical conditions that prohibit general anesthesia. Impossibility of viewing the anatomy adequately. Any situation that, in the doctor's opinion, might involve risk for the patient

* Anticipated difficulty to comply with the investigation (job transfer, geographical distance, lack of motivation, incapacity to fulfill the questionnaires),
* Patient previously included in Robiicca study (for the opposite site)
* Perimodiolar implants (not compatible with the RobOtol®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Speech discrimination score | 1 year
  the speech discrimination score is the percentage of repeated words in silence, with a monosyllabic list, at 60dB, cochlear implant activated.

SECONDARY OUTCOMES:
Speech discrimination score | Baseline, 6 months
  Speech discrimination score (percent of words recognized in monosyllabic list) at 60 dB
Speech Reception Threshold (SRT 50) | 6 months, 12 months
  The speech recognition threshold (SRT) examines at which level 50% of the speech material (usually numbers or spondaic words) is repeated correctly. In addition, SRT gives an index of the hearing sensitivity of speech and helps determine the starting point for other supra-threshold measures such as WR (Word Recognition).
Speech audiometry in noise | 6 months, 12 months
  Signal to Noise Ratio to achieve 50% or 80% intelligibility (SNR50 and SNR80) with the Fra-Matrix noise test
Rate of incomplete insertion | Day one post operative
  Number of electrodes inserted at immediate post-operative imaging by Cone Beam or CT scan.
Rate of electrode translocations | Day one post operative
  Analysis of translocations using software measures after Cone beam or CT scan (blinded centralized analysis)
Residual hearing | Baseline, 6 months, 12 months
  Pure Tone Audiometry thresholds, implant deactivated, at 250, 500, 1000, 2000 and 4000 Hz (mean of the 5 frequencies)
Pure-tone audiometry | 6 months, 12 months
  Pure Tone Audiometry thresholds, implant activated, at 250, 500, 1000, 2000 and 4000 Hz (mean of the 5 frequencies)
Complications related to the implant | Day one, 1 month, 3 months, 6 months, 12 months
  Complications related to implant surgery (peripheral facial palsy, cerebrospinal fluid leaks, neurovegetative disorders, major bleeding, neurological complications, infections, scars disorders, pain, hematoma, dizziness, tinnitus, tympanic perforations, and implant-linked complications : breakdowns, electrode displacements, magnet displacement, implant body displacement, electrode misplaced)
Quality of life of patients with HUI3 | Baseline, one month, 3 months, 6 months, 12 months
  HUI-3 classification system consists of 8 attributes including vision, hearing, speech, ambulation, dexterity, emotion, cognition, and pain. These attributes range from five or six levels of health states for each attribute.
Quality of life of patients with EQ-5D | Baseline, one month, 3 months, 6 months, 12 months
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition.
Vestibular function with VHIT | Baseline, 12 months
  Video head impulse test (vHIT) allows to identify the overt and covert saccades and studies the gain of vestibulo-ocular reflex (VOR) of each semicircular canal.
Vestibular function with Caloric test results | Baseline, 12 months
  The caloric test uses a nonphysiologic stimulus to induce endolymphatic flow in the horizontal semicircular canal and horizontal nystagmus by creating a temperature gradient from one side of the canal to the other.
Vestibular function with MVEP | Baseline, 12 months
  Myogenic Vestibular Evoked Potential (MVEP) detects the presence of reproductible waveforms of normal morphology in latency and amplitude
Incremental cost-effectiveness ratio (cost per point of speech discrimination score gain) from a collective perspective | 12 months
  Effectiveness criteria will be the speech discrimination score (number of words recognized in monosyllabic list) at 60 dB at M12.
  Costs will be estimated in 3 steps: 1) direct costs related to treatment (DRG, length of stay) and one month outpatient resources consumption after surgery; 2) monetary valuation of resources consumed (using NHI official tariffs, and data from the French National Hospitals' Cost Study); 3) cost calculation by multiplying quantities of resources with their corresponding units costs.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MICHEL, Principal Investigator — Nantes University Hospital
Locations (14):
- France (14):
  - Lille University Hospital, Lille, Nord
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Chu Clermont Ferrand, Clermont-Ferrand
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - AP-HM, Marseille
  - CHRU de Montpellier, Montpellier
  - Michel, Nantes
  - CHU NICE, Nice
  - AP-HP - la Pitié-Salpétrière, Paris
  - C.H.R. Pontchaillou, Rennes
  - CHU de Saint-Etienne, Saint-Etienne
  - CHRU Hautepierre, Strasbourg
  - CHRU de Tours, Tours